CLINICAL TRIAL: NCT05227300
Title: Buffered vs. Unbuffered Local Anesthesia in Mandibular Molars Diagnosed With Symptomatic Irreversible Pulpitis: A Controlled, Randomized Double-blind Study
Brief Title: Buffered vs. Unbuffered Local Anesthesia in Mandibular Molars Diagnosed With Symptomatic Irreversible Pulpitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kenneth J. Spolnik DDS, Department of Endodontics Chair, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11447
Record Dates: First submitted 2022-01-07; First posted 2022-02-07 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Symptomatic Irreversible Pulpitis
Keywords: lidocaine; buffered; local anesthetic; irreversible pulpitis
MeSH Terms: interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Intervention Model Description: This study will be a single-center, controlled, randomized, double-blind (provider and subject), 2 treatment, 1 period, parallel study
Who Masked: Participant, Care Provider, Investigator
Masking Description: A statistician will provide a two-product randomization scheme which will randomize each of the 40 subjects on the order of their entry into the study. The research assistants will be aware of and document this scheme, but the student researcher/PI will not know what type of anesthetic will be administered.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Buffered 2% lidocaine with 1:100,000 epinephrine (Experimental): Buffered local anesthetic (addition of sodium bicarbonate to make a 10% buffered solution)
  Interventions: Drug: Onset Sodium Bicarbonate Inj., 8.4%, USP Neutralizing Additive Solution; Drug: 2% lidocaine with 1:100,000 epinephrine
- Unbuffered 2% lidocaine with 1:100,000 epinephrine (Active Comparator): Standard local anesthetic
  Interventions: Drug: 2% lidocaine with 1:100,000 epinephrine

INTERVENTIONS:
Drug: Onset Sodium Bicarbonate Inj., 8.4%, USP Neutralizing Additive Solution — Onpharma's Onset sodium bicarbonate buffer to be added to a standard cartridge of dental local anesthetic
  Arms: Buffered 2% lidocaine with 1:100,000 epinephrine
Drug: 2% lidocaine with 1:100,000 epinephrine — Septodont's standard formulation of 2% lidocaine with epinephrine

SUMMARY:
The purpose of this study is to determine whether one type of anesthetic (numbing medicine) will work better at numbing the nerve in a tooth than using a different type of anesthetic. A second purpose is to see if the time needed to numb the nerve in a tooth is different between the two anesthetics.

DETAILED DESCRIPTION:
40 subjects with a mandibular molar diagnosed with symptomatic irreversible pulpitis will be randomly allocated into 2 groups. One group will receive a total of 3 cartridges of a standard, unbuffered 2% lidocaine with 1:100,000 epinephrine via inferior alveolar nerve block (IANB) followed by supplemental buccal and lingual infiltrations, while the other will receive the equivalent yet buffered formulation. An electronic pulp tester (EPT) will be used to objectively determine baseline pulpal status of the affected tooth, followed by 2-minute interval testing following the administration of all local anesthesia. The onset of pulpal anesthesia is defined by the first of 2 consecutive EPT=80 readings, and the endodontic treatment may begin. Profound pulpal anesthesia is ultimately determined if the patients report a comfortable pulpotomy as reflected on the Wong-Baker FACES Visual Analog Scale.

ELIGIBILITY:
Inclusion Criteria - In order to participate, subjects must:

* Be between the ages of 18 and 80 years old
* Have the ability and willingness to independently consent to treatment and study participation
* Have an uncomplicated medical history (ASA I and II)
* Not be pregnant
* Have no allergies local anesthetics/sulfites (confirmed or self-reported)
* Not be taking any medications that may affect the proper assessment of the anesthetic (no acetaminophen or short-acting NSAIDs such as ibuprofen within the previous 6 hours; no long-acting NSAIDs such as naproxen within the previous 16 hours)
* Not require nitrous oxide during treatment, and the injection area should appear healthy with no other pre-existing conditions or infections that may compromise an accurate collection of data
* Be experiencing signs of irreversible pulpitis (an exaggerated response to cold that lingers longer than 10 seconds) in a mandibular molar at the time of conducting the study

Exclusion Criteria - No subjects will have:

* A negative response to cold in the proposed treatment tooth
* A radiographic periradicular pathosis more advanced than a widened periodontal ligament or have an intraoral swelling

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Dentistry Graduate Endodontics Dept., Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenberg PA, Amin KG, Zibari Y, Lin LM. Comparison of 4% articaine with 1:100,000 epinephrine and 2% lidocaine with 1:100,000 epinephrine when used as a supplemental anesthetic. J Endod. 2007 Apr;33(4):403-5. doi: 10.1016/j.joen.2006.11.019. Epub 2007 Feb 20. PMID 17368327
- [Background] Goodis HE, Poon A, Hargreaves KM. Tissue pH and temperature regulate pulpal nociceptors. J Dent Res. 2006 Nov;85(11):1046-9. doi: 10.1177/154405910608501114. PMID 17062748
- [Background] Christoph RA, Buchanan L, Begalla K, Schwartz S. Pain reduction in local anesthetic administration through pH buffering. Ann Emerg Med. 1988 Feb;17(2):117-20. doi: 10.1016/s0196-0644(88)80293-2. PMID 2827545
- [Background] Schellenberg J, Drum M, Reader A, Nusstein J, Fowler S, Beck M. Effect of Buffered 4% Lidocaine on the Success of the Inferior Alveolar Nerve Block in Patients with Symptomatic Irreversible Pulpitis: A Prospective, Randomized, Double-blind Study. J Endod. 2015 Jun;41(6):791-6. doi: 10.1016/j.joen.2015.02.022. Epub 2015 Apr 1. PMID 25841959
- [Background] Saatchi M, Farhad AR, Shenasa N, Haghighi SK. Effect of Sodium Bicarbonate Buccal Infiltration on the Success of Inferior Alveolar Nerve Block in Mandibular First Molars with Symptomatic Irreversible Pulpitis: A Prospective, Randomized Double-blind Study. J Endod. 2016 Oct;42(10):1458-61. doi: 10.1016/j.joen.2016.07.004. Epub 2016 Aug 6. PMID 27507627
- [Background] Fowler S, Reader A. Is a volume of 3.6 mL better than 1.8 mL for inferior alveolar nerve blocks in patients with symptomatic irreversible pulpitis? J Endod. 2013 Aug;39(8):970-2. doi: 10.1016/j.joen.2013.04.007. Epub 2013 May 16. PMID 23880260
- [Background] Kanaa MD, Whitworth JM, Meechan JG. A prospective randomized trial of different supplementary local anesthetic techniques after failure of inferior alveolar nerve block in patients with irreversible pulpitis in mandibular teeth. J Endod. 2012 Apr;38(4):421-5. doi: 10.1016/j.joen.2011.12.006. Epub 2012 Feb 2. PMID 22414822

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Buffered 2% Lidocaine With 1:100,000 Epinephrine | Unbuffered 2% Lidocaine With 1:100,000 Epinephrine
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients present with signs of symptomatic irreversible pulpitis on a mandibular molar.
Groups:
- Total: Total of all reporting groups
Arm/Group | Buffered 2% Lidocaine With 1:100,000 Epinephrine | Unbuffered 2% Lidocaine With 1:100,000 Epinephrine | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.2 (13.5) | 38 (19.4) | 39.6 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 23
  Male | 5 | 12 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Initial Visual Analog Scale (VAS) w/ a min score of 1 and max score of 10 (a 4+ is significant pain) [Mean (Full Range); unit: Units on a Scale] — The Visual Analog Scale used in this study ranges from a minimum of 1 (no pain) to a maximum score of 10 (most extreme pain). A VAS score of 4 is considered to be the lower end of moderate pain which is categorized as significant in our study. Therefore, a recorded initial VAS of 4 or greater constitutes a symptomatic irreversible pulpitis and qualifies for our study.
  Units on a Scale | 7.8 [4 to 10] | 6.9 [5 to 10] | 7.35 [4 to 10]
Initial Electronic Pulp Test (EPT) less than 80 shows vital pulp (min stimulation is 1, max is 80) [Mean (Full Range); unit: Units on a scale] — If an initial EPT test reflects any score under 80 (1-79), then there is evidence of vital pulpal tissue that is necessary to be included in our study. An initial EPT score of 80 demonstrates necrotic pulpal tissue since there is no sensory nerve conduction present to start and the patient would not qualify for the study. Also to note- after successful anesthesia the EPT would reflect a score of 80 because the anesthesia blocks the sensory nerve conduction.
  Units on a scale | 42.9 [30 to 71] | 47.3 [14 to 72] | 45.1 [14 to 72]

OUTCOME MEASURES:

1. Primary Outcome: VAS Scores as Measures of Profoundness of Pulpal Anesthesia
Description: The mean Visual Analog Scale (VAS) score, which ranges from a min of 1 to a max of 10. In other words, inadequate anesthesia is considered to be a VAS score that is between 4 and 10 because that is not considered to be "comfortable and profound".
Time Frame: Up to 20 minutes post-drug administration
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Buffered 2% Lidocaine With 1:100,000 Epinephrine | Unbuffered 2% Lidocaine With 1:100,000 Epinephrine
Number analyzed (Participants) | 20 | 20
Score on a scale | 3.1 [0 to 8] | 1.2 [0.0 to 7]

2. Secondary Outcome: Onset of Pulpal Anesthesia
Description: Duration of time in minutes required to achieve pulpal anesthesia, defined as an electrical pulp test score of 80 (which is the maximum stimulation). Any EPT score between 1-79 after 20 minutes post-anesthesia is considered a failure of pulpal anesthesia.
Time Frame: Up to 20 minutes post-drug administration
Measure: Mean (Full Range); unit: Minutes
Arm/Group | Buffered 2% Lidocaine With 1:100,000 Epinephrine | Unbuffered 2% Lidocaine With 1:100,000 Epinephrine
Number analyzed (Participants) | 20 | 20
Minutes | 8.4 [3.8 to 14] | 8.8 [3.2 to 17.2]

ADVERSE EVENTS:
Time Frame: 3.5 month enrollment period; each patient's data was collected at a single treatment appointment within the specified enrollment period; each of these appointments last on average 3 hours.
Description: Adverse event is defined as a negative event that is outside the typical possible reaction that a patient could routinely experience while undergoing dental local anesthesia at a single dental appointment.
Arm/Group | Buffered 2% Lidocaine With 1:100,000 Epinephrine | Unbuffered 2% Lidocaine With 1:100,000 Epinephrine
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
With a total sample size of 40 (20 subjects per group), this study has an 80% power to detect a difference between 90% and 50% of subjects who achieve profound pulpal anesthesia. Increasing the sample size to include a larger number of subjects per group would also increase the power and ultimately the level of statistical significance between those groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT05227300/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT05227300/ICF_000.pdf